CLINICAL TRIAL: NCT00097279
Title: A Multicenter, Open-Label, Randomised Trial to Compare the Efficacy and Safety of NovoLog Mix 70/30 BID in Combination With Metformin and Pioglitazone to Metformin and Pioglitazone Alone in Insulin Naïve Subjects With Type 2 Diabetes
Brief Title: Comparison of Biphasic Insulin Aspart 70/30 With Anti-Diabetic Drugs in Subjects With Type 2 Diabetes
Acronym: ACTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-2186
Record Dates: First submitted 2004-11-19; First posted 2004-11-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Pioglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: pioglitazone
Drug: metformin

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this study is to test whether biphasic insulin aspart 70/30 is a safe and at least as effective alternative in combination with two oral anti-diabetics compared to the two oral anti-diabetics alone for the control of blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2004-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 24 weeks

SECONDARY OUTCOMES:
Safety variables
Other glycemic variables
8-point plasma glucose profiles

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (70):
- United States (70):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Burlingame, California
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Redwood City, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, New Britain, Connecticut
  - Novo Nordisk Investigational Site, Newark, Delaware
  - Novo Nordisk Investigational Site, Aventura, Florida
  - Novo Nordisk Investigational Site, Fort Myers, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Easton, Maryland
  - Novo Nordisk Investigational Site, Danvers, Massachusetts
  - Novo Nordisk Investigational Site, Salisbury, Massachusetts
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Grand Rapids, Michigan
  - Novo Nordisk Investigational Site, Livonia, Michigan
  - Novo Nordisk Investigational Site, Saint Cloud, Minnesota
  - Novo Nordisk Investigational Site, Columbia, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Reno, Nevada
  - Novo Nordisk Investigational Site, Hampton, New Hampshire
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Turnersville, New Jersey
  - Novo Nordisk Investigational Site, East Syracuse, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Medford, Oregon
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Suffolk, Virginia
  - Novo Nordisk Investigational Site, Warrenton, Virginia
  - Novo Nordisk Investigational Site, Kirkland, Washington
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Raskin P, Matfin G, Schwartz SL, Chaykin L, Chu PL, Braceras R, Wynne A. Addition of biphasic insulin aspart 30 to optimized metformin and pioglitazone treatment of type 2 diabetes mellitus: The ACTION Study (Achieving Control Through Insulin plus Oral ageNts). Diabetes Obes Metab. 2009 Jan;11(1):27-32. doi: 10.1111/j.1463-1326.2007.00796.x. Epub 2007 Oct 17. PMID 17941873
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com